CLINICAL TRIAL: NCT00775034
Title: Drainage Versus Sealant in Double Blinded Monocentric Open Incisional Hernia Repair
Acronym: DREAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008/433
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia | interventions — Fibrin Tissue Adhesive; Drainage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Study group (Tisseel®)
  Interventions: Drug: Tisseel®
- 2 (Other): Control group
  Interventions: Procedure: Drainage

INTERVENTIONS:
Drug: Tisseel® — Mesh repair for open incisional hernia repair with fibrin sealant
  Arms: 1
Procedure: Drainage — Mesh repair for open incisional hernia repair with drainage
  Arms: 2

SUMMARY:
Mesh repair for open incisional hernia repair with fibrin sealant or with drainage

ELIGIBILITY:
Inclusion Criteria:

* All patients with a large incisional hernia >5cm diameter that needs elective repair with mesh augmentation

Exclusion Criteria:

* no written informed consent
* 'hostile' abdomen
* emergency surgery (incarcerated hernia)
* parastomal hernia
* incisional hernia outside the midline
* recurrent incisional hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-01-27 (Actual); Primary Completion 2014-10-14 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Hospital stay | At time of discharge

SECONDARY OUTCOMES:
Postoperative drainage volume | Day 0,1, 2, 3 ? and at day of removal
Perioperative morbidity rate | At time of discharge
Pain measured using VAS | Daily till discharge and after 3 weeks post-surgery
Quality of life by SF-36 questionnaire | Preoperatively, at time of discharge, 2 weeks after discharge, 6 weeks after discharge and 1 year post surgery
Recurrence | At one year

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - University Hospital Ghent, Ghent
  - UZ gasthuisberg Leuven, Leuven

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be